CLINICAL TRIAL: NCT00765765
Title: Phase I/II Study of Ixabepilone in Combination With the Autophagy Inhibitor Hydroxychloroquine for the Treatment of Patients With Metastatic Breast Cancer
Brief Title: Ixabepilone and Hydroxychloroquine in Treating Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000615000; P30CA072720 (NIH); CINJ-040804 (Other: CINJ); 0220080205 (Other: Rutgers University IRB)
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2023-08-09 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Hydroxychloroquine; ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ixabepilone and hydroxychloroquine (Experimental)
  Interventions: Drug: hydroxychloroquine; Drug: ixabepilone

INTERVENTIONS:
Drug: hydroxychloroquine — Dose escalation from 200 mg po qd to 200 mg po bid.
Drug: ixabepilone — Starting dose of 40 mg/m2 and can dose reduce to 32 mg/m2.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ixabepilone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Hydroxychloroquine may help ixabepilone work better by making tumor cells more sensitive to the drug.

PURPOSE: This phase I/II trial is studying the side effects and best dose of ixabepilone given together with hydroxychloroquine and to see how well they work in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* The primary objective of this study is to assess the antitumor activity, measured by tumor response rate, in patients who receive this regimen as a third-line treatment. (Phase II)

Secondary

* To measure the duration of response for responding patients.
* To measure the time to progressive disease.
* To measure survival time.
* To characterize the quantitative and qualitative toxicities of this regimen in these patients.
* To develop pharmacodynamic markers for autophagy detection in patient specimens.
* To characterize the effects of hydroxychloroquine on autophagy in patients in vivo.
* To investigate whether the estrogen receptor, progesterone receptor, and/or HER2 status of breast tumors correlates with treatment response.

OUTLINE: This is a multicenter, phase I dose-escalation study of ixabepilone followed by a phase II study.

During the first course, patients receive ixabepilone IV over 3 hours on day 1 and oral hydroxychloroquine twice daily on days 3-21. On all subsequent courses, patients receive ixabepilone IV over 3 hours on day 1 and oral hydroxychloroquine twice daily on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Histologic or cytologic elements can be established on metastatic tumor aspirate or biopsy
  * Metastatic disease
  * Measurable disease according to RECIST criteria
* Must have received 2 prior chemotherapy regimens for metastatic breast cancer
* Anthracycline-resistant (or treated with minimum cumulative doxorubicin dose of 240 mg/m^2 or epirubicin dose of 360 mg/m^2) and taxane-resistant disease

  * Anthracycline resistance is defined as progression while on therapy or within 6 months in the adjuvant/neoadjuvant setting or 3 months in the metastatic setting
  * Taxane resistance is defined as progression while on therapy or within 12 months in the adjuvant/neoadjuvant setting or 4 months in the metastatic setting
* Hormone receptor status known
* No known CNS metastases or previously treated and now stable CNS metastases

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-2
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ upper limit of normal (ULN)

  * If patient has Gilbert's disease, then patient must have isolated hyperbilirubinemia (e.g., no other liver function test abnormality), with maximum bilirubin ≤ 2 times ULN
* AST and ALT ≤ 2.5 times ULN, independently of liver metastases
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN OR calculated creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other active malignancy

  * History of basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix within the past 3 years allowed provided patient has been treated with curative intent
  * History of prior malignancy allowed provided patient has been treated with curative intent and has been disease free > 3 years
* None of the following conditions within the past 6 months:

  * Myocardial infarction
  * Stroke
  * Symptomatic peripheral vascular disease
* No unstable angina or NYHA class II-IV congestive heart failure
* No history of psoriasis or porphyria
* No history of hypersensitivity to 4-aminoquinoline compound
* No retinal or visual field changes from prior 4-aminoquinoline-compound use
* No history of G6PD deficiency
* No GI pathology that would interfere with drug bioavailability
* No motor or sensory neuropathy ≥ grade 2 (NCI CTCAE) at study entry
* No serious uncontrolled medical disorder or active infection at study entry
* No rheumatoid arthritis or systemic lupus erythematosus requiring active treatment
* No history of HIV
* No history of any condition (social or medical) that, in the opinion of the investigator, might interfere with the patient's ability to comply with the protocol or pose additional or unacceptable risk to the patient

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior radiation to tumor sites allowed provided:

  * Radiation was completed ≥ 3 weeks prior to study treatment
  * All radiation-related toxicities have resolved to ≤ grade 1
* No more than 3 prior chemotherapy regimens in the metastatic setting
* No prior ixabepilone or another epothilone
* No concurrent highly active antiretroviral therapy
* No other concurrent hydroxychloroquine for treatment or prophylaxis of malaria
* No other concurrent anticancer investigational or commercial agents or therapies

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vassil Karantza-Wadsworth, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/show/NCT00765765

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six subjects were recruited from The Cancer Institute of New Jersey (a comprehensive cancer center) and one of its affiliate community hospitals in New Jersey, from April 2009 through June 2010.
Groups:
- Ixabepilone and Hydroxychloroquine: ixabepilone : Starting dose of 40 mg/m2 and can dose reduce to 32 mg/m2.
  hydroxychloroquine : Dose escalation from 200 mg po qd to 200 mg po bid.
Period: Overall Study
Arm/Group | Ixabepilone and Hydroxychloroquine
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ixabepilone and Hydroxychloroquine
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Secondary Outcome: Duration of Response
Time Frame: 5 years
Population: The study was closed early due to slow accrual. Insufficient data were collected to analyze this outcome measure.
Arm/Group | Ixabepilone and Hydroxychloroquine
Number analyzed (Participants) | 0

2. Secondary Outcome: Time to Progressive Disease
Time Frame: 5 years
Population: The study was closed early due to slow accrual. Insufficient data were collected to analyze this outcome measure.
Arm/Group | Ixabepilone and Hydroxychloroquine
Number analyzed (Participants) | 0

3. Secondary Outcome: Survival Time
Time Frame: 5 years
Population: The study was closed early due to slow accrual. Insufficient data were collected to analyze this outcome measure.
Arm/Group | Ixabepilone and Hydroxychloroquine
Number analyzed (Participants) | 0

4. Secondary Outcome: Pharmacodynamic Markers for Autophagy Detection
Time Frame: 2 years
Population: The study was closed early due to slow accrual. Insufficient data were collected to analyze this outcome measure.
Arm/Group | Ixabepilone and Hydroxychloroquine
Number analyzed (Participants) | 0

5. Secondary Outcome: Effects of Hydroxychloroquine on Autophagy
Time Frame: 2 years
Population: The study was closed early due to slow accrual. Insufficient data were collected to analyze this outcome measure.
Arm/Group | Ixabepilone and Hydroxychloroquine
Number analyzed (Participants) | 0

6. Secondary Outcome: Correlation of Estrogen Receptor, Progesterone Receptor and/or HER2 Status With Treatment Response
Time Frame: 5 years
Population: The study was closed early due to slow accrual. Insufficient data were collected to analyze this outcome measure.
Arm/Group | Ixabepilone and Hydroxychloroquine
Number analyzed (Participants) | 0

7. Primary Outcome: Tumor Response Rate
Description: Overall Complete Response and Partial Response will be considered tumor response. Ixabepilone as a single agent (40 mg/m2 as an intravenous infusion every 3 weeks) was evaluated in a previous (Phase II) study in women with metastatic breast cancer and that the objective tumor response rate was 11.5%. In another(Phase III) study, Ixabepilone in combination with capecitabine resulted in an objective tumor response rate of 35%, compared to that of capecitabine alone (14%). Therefore, in the Phase II portion of the ixabepilone plus hydroxychloroquine combination treatment study, a tumor response rate of less than 15% will be deemed uninteresting. The target tumor response rate will be 35%. Due to uncertainty about the true response rate of ixabepilone plus hydroxychloroquine combination on this patient poupation, we also will consider a response rate of 30% to be encouraging.
Time Frame: 3 years
Population: The study was closed early due to slow accrual. Insufficient data were collected to evaluate this outcome measure.
Arm/Group | Ixabepilone and Hydroxychloroquine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Arm/Group | Ixabepilone and Hydroxychloroquine
All-Cause Mortality (participants affected / at risk) | 6/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixabepilone and Hydroxychloroquine (N=6)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixabepilone and Hydroxychloroquine (N=6)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4 (15)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3 (7)
Blood/Bone Marrow (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Pain - Abdomen NOS (General disorders) | 1 (1)
Pain - Back (General disorders) | 1 (1)
Pain - Bone (General disorders) | 1 (1)
Pain - Chest wall (General disorders) | 1 (1)
Pain - Joint (General disorders) | 1 (1)
Pain - Muscle (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cardiac General (Cardiac disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory - Nose (Vascular disorders) | 1 (1)
Mood alteration - Depression (Psychiatric disorders) | 1 (1)
Vision-flashing lights/floaters (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes